CLINICAL TRIAL: NCT01731704
Title: A Randomized Controlled Study Of Neurocognitive Outcomes In Patients With Five Or More Brain Metastases Treated With Radiosurgery Or Whole-Brain Radiotherapy
Brief Title: Neurocognitive Outcomes In Patients Treated With Radiotherapy For Five Or More Brain Metastases
Acronym: NAGKC 12-01
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: University of California, San Francisco (Other)
Collaborators: North American Gamma Knife Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121010/12-01
Record Dates: First submitted 2012-11-07; First posted 2012-11-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Brain Metastases
Keywords: 5 or more brain metastases; proven diagnosis of a non-hematopoietic malignancy; non-small cell lung cancer or germ cell malignancy
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stereotactic Radiosurgery (SRS) (Active Comparator): Radiation Therapy: Radiosurgical (SRS) technique via Gamma Knife Perfexion radiosurgical system
  Interventions: Radiation: Stereotactic radiosurgery (SRS)
- Whole Brain Radiation Therapy (WBRT) (Active Comparator): whole-brain radiation therapy 30 Gy in 10 fractions. Treatment will be delivered once daily, 5 fractions per week, over 2 to 2.5 weeks
  Interventions: Radiation: Whole brain radiation therapy (WBRT)

INTERVENTIONS:
Radiation: Stereotactic radiosurgery (SRS)
  Other Names: Gamma knife Perfexion radiosurgical device
  Arms: Stereotactic Radiosurgery (SRS)
Radiation: Whole brain radiation therapy (WBRT) — External beam whole-brain radiation therapy 30 Gy in 10 fractions. Treatment will be delivered once daily, 5 fractions per week, over 2 to 2.5 weeks
  Arms: Whole Brain Radiation Therapy (WBRT)

SUMMARY:
This is randomized study of neurocognitive outcomes in patients with five or more brain metastases treated with stereotactic radiosurgery (SRS), specifically the Gamma Knife (GK) system, or whole-brain radiation therapy (WBRT). The primary aim of this study is to compare the change in neurocognitive function outcome between baseline and 6 months in WBRT versus SRS treatment groups.

DETAILED DESCRIPTION:
This is randomized controlled study of neurocognitive outcomes in patients with five or more brain metastases treated with stereotactic radiosurgery (SRS), specifically the Gamma Knife (GK) system, or whole-brain radiation therapy (WBRT). The goal of the study is to enroll 120 patients with at least five (≥5) newly-diagnosed brain metastases from non-melanoma, except melanoma patients with BRAF V600E B-Raf protein mutation, primary cancers with the largest intracranial tumor volume ≤10 cc, ≤15 cc total tumor volume, absence of leptomeningeal disease on MRI, and Karnofsky performance status (KPS) score ≥70 (unless due to intracranial disease), and KPS expected to improve to ≥70 with treatment.

All study participants will undergo standard, pre-treatment clinical evaluations that include: complete clinical/neurologic exam, performance status assessment, systemic staging, and diagnostic MRI of the brain. The baseline neurocognitive function (NCF) will be assessed by a short (20-30 minute) online test battery that can be completed by patients at home. All study participants will be randomized to receive radiosurgical or whole-brain radiation treatment for their brain metastases. All patients will have treatment response assessments every 10-12 weeks consisting of a clinical/neurologic exam, performance status evaluation, disease re-staging (if indicated), and diagnostic MRI of the brain. If progressive disease is identified (radiographic progression of treated lesions or new brain lesions), the patients will be considered for "salvage" therapy which will primarily consist of SRS, WBRT, surgery±brachytherapy or best supportive care (e.g. steroids only). The preferred salvage therapy will be SRS provided that the re-treatment criteria are met. The NCF follow-up will start 2 weeks after completion of the initial SRS treatment and will repeat at 2-week intervals, irrespective of any salvage therapy that may be indicated. All study participants will be followed until death or withdrawal from the study.

The primary aim of this study is to compare the change in neurocognitive outcome between baseline and 6 months for surviving patients in upfront WBRT versus SRS treatment groups. The primary study endpoint is neurocognitive function as measured by a significant change in online neurocognitive function (oNCF) z-score from baseline to 6 months. The outcomes will be compared after initial treatment and then repeatedly in follow-up, and will include the impact of salvage SRS treatments. This approach will allow us to assess the relative impact on neurocognitive outcomes of repeat SRS treatments to sites of new brain metastases.

Since SRS and WBRT are two very different forms of treatment (single high-dose treatment vs. multiple low-dose treatments) with markedly different target volumes, it is expected that local control rates will also be markedly different. This, in turn, will impact salvage therapies and associated costs. This study will evaluate local control rates and overall intracranial disease control at 3, 6, 9, and 12 months as a function of initial treatment cohort (SRS vs. WBRT). We also expect significant differences between the treatment groups in patient and caregiver reported quality of life (QoL) measures.

It is also expected that the SRS cohort will require multiple SRS treatments over the course of the study since, unlike WBRT, the treatments target only gross brain metastases and do not address microscopic (clinically undetectable) disease. Conversely, WBRT is expected to result in inferior control rates of gross metastatic disease, increasing the likelihood of subsequent SRS or other salvage therapy. For these reasons, we will track the actual costs of treatments over the course of the study, including the need for supportive care and the ability of patients to continue to work in their previous occupation.

The structure of the current study provides a unique opportunity to explore various dosimetric SRS parameters in the setting of multiple brain metastases. Dose-volume criteria for SRS have been established in a prospective RTOG 90-05 dose-finding study and subsequently validated in RTOG 95-08, a randomized controlled trial of WBRT±SRS in patients with 1-3 brain metastases. Several single-institution series as well as multi-institutional retrospective analyses support the use of single-dose SRS for treatment of brain metastases; however, the dose-volume criteria and prescription guidelines are not known in the setting of ≥5 brain metastases where dose interaction among different lesion targets are much more likely. These interactions can potentially lead to increased rates of radiation necrosis, and if the SRS doses are arbitrarily reduced because of such concerns, then to a potentially decreased local control rates. These parameters will be closely tracked in this study with the aim of establishing an evidence-based dosimetric guidelines for radiosurgical treatment of multiple (≥5) brain metastases.

The data gained from this study could help define patient selection and treatment criteria for SRS of multiple brain metastases as a potential alternative to WBRT in a select group of patients. This will also be a first study of its kind to use online neurocognitive assessments for its primary endpoints to demonstrate feasibility and cost-effectiveness of such an approach in a multi-institutional setting.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of a non-hematopoietic malignancy other than small cell lung cancer and germ cell malignancy within 5 years of registration. If the original histologic proof of malignancy is greater than 5 years, then pathological confirmation is required (e.g. from extra- or intra-cranial disease).
* If an open biopsy is performed, the patient must be at least one week post biopsy. This requirement does not apply to patients who undergo stereotactic biopsies.
* Patients with ≥5 measurable brain metastases on a diagnostic-quality contrast-enhanced magnetic resonance imaging (MRI) obtained within 30 days prior to registration.
* Patients with ≤10 cc largest tumor volume, and ≤15 cc total tumor volume.
* History/physical examination within 30 days prior to registration.
* Age ≥18 years.
* Karnofsky performance status ≥70 (RTOG recursive partitioning analysis (RPA) Class I & II).
* Minimum pre-treatment oNCF score ≥70.
* Patients must provide study-specific informed consent prior to study entry.
* Women of child-bearing age must have a negative, quantitative serum pregnancy test ≤14 days prior to study entry, or have a documented reason why such a test is not necessary (e.g. history of tubal ligation).
* Patients must be able to speak and read English fluently (required for the use of online NCF testing).
* Patients must demonstrate basic computer literacy skills and have access to an internet terminal (required for the use of online NCF testing).

Exclusion Criteria:

* Clinical (e.g. multiple new cranial nerve deficits in the absence of obvious radiographic disease to explain symptoms) or radiographic evidence of leptomeningeal disease.
* Patients with measurable brain metastasis(es) resulting from small cell lung cancer and/or germ cell malignancy.
* No documentation of prior cytotoxic or other therapy for malignancy if such therapy was previously received. Note: This does not apply to patients with synchronous metastases at initial diagnosis.
* Contraindication to MR imaging, such as implanted metal devices or foreign bodies, severe claustrophobia, or contraindications to contrast agent administration.
* Estimated glomerular filtration rate (eGFR) <60 within 6 weeks prior to registration. • Prior radiation therapy to the brain. • Severe, active co-morbidity, defined as follows:

  * Unstable angina, and/or congestive heart failure requiring hospitalization within the last 6 months.
  * Transmural myocardial infarction within the last 6 months. - Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization, or precluding study therapy at the time of registration.
  * Uncontrolled, clinically significant cardiac arrhythmias. - Radiologic or clinical evidence of hydrocephalus, or history of previously treated hydrocephalus.
* Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study is potentially teratogenic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10-26 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
To compare the relative change in neurocognitive outcomes (change in oNCF z-score) between baseline and 6 months for surviving patients in upfront WBRT vs. SRS treatment groups. | Every 3 months for 12 months
  All participants will be asked to complete:
  1. Online brain function testing: Complete a short 20-minute online brain function (cognitive) assessment every 2 weeks (twice per month, at least 10-14 days apart).
  2. Quality of Life Questionnaire: Complete a self-reported (if patient) and caregiver quality of life questionnaires every 10-12 weeks (2.5-3 months). These questionnaires take approximately 15-20 minutes to complete and can be done online or in clinic during follow-up visits.

SECONDARY OUTCOMES:
To compare the relative change in neurocognitive outcomes (change in oNCF z-score) between baseline and 12 months for surviving patients in upfront WBRT vs. SRS treatment groups. | Every 10-12 weeks for 12 months after treatment
  * Neurocognitive function, 12-months post whole-brain radiation therapy (WBRT)/stereotactic radiosurgery (SRS)specifically the Gamma Knife (GK) system, treatment as measured by the online neurocognitive function (oNCF) composite z-score.
  * Neurocognitive function at all time points as measured by the online neurocognitive function (oNCF) composite z-score.
To compare the relative impact of initial therapy on patients' quality of life (QoL) as measured by caregiver assessments | Every 10-12 weeks for 12 months after treatment
  • Quality of life (patient-reported measures) as measured by Beck Depression Inventory, Beck Anxiety Inventory, FACT-Br, FACT-Cog, Fatigue Severity Scale, EuroQol(EQ5D), EORTC-BN20, and QOL-30.
To compare the relative impact of initial therapy on patients' quality of life (QoL) as measured by caregiver assessments | Every 10-12 months
  Quality of life as measured by caregiver assessments including Frontal Systems Behavior Scale, Neuropsychiatric Inventory, Functional Activities Questionnaire, and Everyday Cognition Questionnaire.
To estimate consistency and change in z-scores for oNCF assessments over all study endpoints in surviving patients treated with upfront whole brain radiation therapy (WBRT) vs. stereotactic radiosurgery (SRS). | Every 10-12 months
To compare proportions of patients in the two treatment groups that require salvage therapy as a function of systemic disease control (controlled vs. uncontrolled). | 3, 6, 9, and 12 months
To compare the overall survival between patients in upfront whole brain radiation therapy (WBRT) vs. stereotactic radiosurgery (SRS) treatment groups | baseline to study completion

OTHER OUTCOMES:
Cost analysis | Prior to treatment up to 12 months after treatment is complete
  To determine what healthcare cost data can be collected in patients with metastatic disease within a context of a multi-institutional clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Igor J Barani, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States